CLINICAL TRIAL: NCT01469078
Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered as Single Bolus Injections in Subjects With Stage 5 Chronic Kidney Disease on Dialysis Therapy (CKD-5D) (PK-CKD-05)
Brief Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered as Single Bolus Injections in Subjects With Stage 5 Chronic Kidney Disease on Dialysis Therapy (CKD-5D)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Collaborators: ClinSmart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: P-Monofer-PK-CKD-05
Record Dates: First submitted 2011-10-27; First posted 2011-11-10 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic Kidney Disease; CKD stage 5; Iron deficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Iron Deficiencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 100 mg Monofer® (Active Comparator)
  Interventions: Drug: Monofer®
- 200 mg Monofer® (Active Comparator)
  Interventions: Drug: Monofer®
- 500 mg Monofer® (Active Comparator)
  Interventions: Drug: Monofer®

INTERVENTIONS:
Drug: Monofer® — Single Bolus Injections

SUMMARY:
The purpose of this study is to assess Pharmakokinetic properties of iron isomaltoside 1000 (Monofer®) in doses of 100 mg, 200 mg or 500 mg in subjects with Stage 5 Chronic Kidney Disease on Dialysis Therapy (CKD-5D).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Weight above 50 kg.
3. Subjects diagnosed with CKD-5D and on dialysis therapy for at least 90 days prior to inclusion.
4. Serum ferritin ≤ 800 ng/mL.
5. Transferrin Saturation ≤ 35%.
6. Life expectancy beyond 12 months by Principal Investigator's judgement.
7. Hb concentrations ≥10.0 g/dL and ≤12.5 g/dL both at Screening Visit 1a and at Screening Visit 1b (Screening Visit 1a and Visit 1b must be separated by at least 1 week).
8. Erythropoiesis Stimulating Agent (ESA) treatment (to be kept constant during the study period and for 4 weeks prior to inclusion with only one missed dose to be allowed during this pre-entry period).
9. Subjects in maintenance iron therapy with average iron administration ≤ 100 mg/week for 4 weeks prior to inclusion and willingness to switch to investigational product.
10. Willingness and ability to participate after informed consent (including HIPAA, if applicable).

Exclusion Criteria:

1. Anemia caused primarily by other factors than renal related anemia.
2. Iron overload or disturbances in utilization of iron (e.g. hemochromatosis and hemosiderosis).
3. Difference of Hb ≥ 1.0 g/dL between Screening Visits 1a and 1b.
4. Known hypersensitivity to any excipients in the investigational drug products.
5. Subjects with a history of multiple allergies.
6. Decompensated liver cirrhosis and history of hepatitis B or C [Alanine Aminotransferase (ALT) > 3 times upper limit of normal].
7. Acute or chronic infections (assessed by clinical investigator judgment), supported by White Blood Cells (WBC) and C-Reactive Protein (CRP).
8. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
9. Pregnant or nursing women.
10. Women of child bearing potential who are not using safe contraceptive methods (e.g. intrauterine device, oral contraceptives or surgically sterilized) or who are planning to become pregnant within the study period.
11. Blood transfusion within the previous 12 weeks.
12. Planned elective surgery during the study where significant blood loss is expected.
13. Participation in any other clinical trial within 3 months prior to screening.
14. Untreated Vitamin B12 or folate deficiency.
15. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study. Examples include Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-10; Primary Completion 2012-04 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Determination of changes in Iron pharmacokinetic parameters from plasma/serum concentration profile | From exposure to 7 days post-exposure
  The follwoing parameter will be determined: AUC0-t, AUC, Cmax, Tmax, Ke, and T1/2

SECONDARY OUTCOMES:
Changes in pharmacodynamic parametres | From 0 hours to 4, 8, 24, 48, 72 hours post-exposure and end of study visit
  Changes in the following parametres will be determined: Hemoglobin (Hb), Reticulocyte Count, Reticuloycyte Hemoglobin Content (CHr), Ferritin, Total Iron Binding Capacity (TIBC) and Transferrin Saturation (TfS)
Safety evaluation | From screening to 7 days post-exposure
  The following parameters will be evaluated: Laboratory safety variable, physical examination, vital signs and Electrocardiogram (ECG)